CLINICAL TRIAL: NCT06896409
Title: PuraStat® Combined With Adrenaline Versus Standard of Care in Non-variceal Upper Gastrointestinal Bleeding. Multicentric International Clinical Trial.
Brief Title: PuraStat® Combined With Adrenaline Versus Standard of Care in Upper Gastrointestinal Bleeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tallaght University Hospital (Other)
Responsible Party: Principal Investigator, Raquel Ballester, Principal Investigator, Tallaght University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUR02
Record Dates: First submitted 2025-02-01; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Epinephrine; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PuraStat® combined with Adrenaline (Experimental): In this experimental arm PuraStat® (mL) will be administered in combination with an injection of Adrenaline (mL).
  Interventions: Combination Product: PuraStat® combined with Adrenaline
- Standard of Care (Active Comparator): This arm will be the active comparator, will include all types of standard of care currently recommended for the treatment of bleeding lesions, such as, adrenaline injection + second hemostasis modality (contact thermal, mechanical therapy, or injection of a sclerosing agent).
  Interventions: Combination Product: Standard of Care

INTERVENTIONS:
Combination Product: PuraStat® combined with Adrenaline — PuraStat® application (mL) combined with Adrenaline injection (mL)
  Arms: PuraStat® combined with Adrenaline
Combination Product: Standard of Care — Adrenaline injection + second hemostasis modality (contact thermal, mechanical therapy, or injection of a sclerosing agent).
  Arms: Standard of Care

SUMMARY:
PuraStat® is a novel gel that offers several advantages over traditional hemostatic powders. Its transparency allows for continuous visualization of the bleeding site, and it can be applied in narrow spaces or in combination with other treatments. Additionally, the pre-filled syringe design ensures ease of handling and precise delivery.

Most published data on PuraStat® as a hemostatic agent originates from surgical settings. In endoscopy, its primary applications have been in polypectomy-related hemostasis and the promotion of wound healing. Reports indicate a hemostasis success rate of 90.4%, with a recurrence rate of 10.4%.

Limited data exist regarding the efficacy of PuraStat® as a hemostatic agent in upper gastrointestinal bleeding (UGIB) lesions. This study hypothesizes that PuraStat®, when combined with Adrenaline, serves as a feasible and effective first-line treatment for gastrointestinal bleeding. To evaluate this, a prospective, randomized, parallel-group, open-label clinical trial is proposed.

DETAILED DESCRIPTION:
Endoscopic treatment serves as the first-line approach in managing upper gastrointestinal bleeding (UGIB), demonstrating effectiveness in reducing re-bleeding rates, the need for surgical intervention, and mortality. In non-variceal UGIB, endoscopic management includes various techniques such as injection therapy, thermal therapy, mechanical therapy, or a combination, depending on the lesion type. However, certain factors, including the anatomical location of the lesion, underlying fibrosis, or diffuse bleeding, can present challenges to successful treatment.

Haemostatic powders have been increasingly utilized as both primary and salvage therapy for bleeding control in various clinical scenarios, including post-polypectomy bleeding, bleeding associated with colonic tumors, diverticula, arteriovenous malformations, radiation proctitis, ischemic colitis, and surgical intestinal anastomoses. Their use in UGIB management has also expanded. Compared to other modalities, these topical agents offer advantages such as ease of application, the ability to reach lesions in challenging locations, and coverage of larger surface areas without requiring precise targeting.

Among the most extensively studied topical hemostatic agents are TC-325 (Hemospray®, Cook Medical), the Polysaccharide Hemostatic System (Endoclot® PHS), and Inha University-Endoscopic Wound Dressing (UI-EWD) (NextBiomedical Co., Incheon, South Korea). These agents have demonstrated high rates of immediate haemostasis (86%-100%) when used alone or in combination with other haemostatic methods, exhibiting excellent feasibility and a favorable safety profile.

The primary limitation of these agents is their adherence exclusively to actively bleeding sites, leading to rapid washout within 12-24 hours, thereby making them a temporary measure. Additionally, their opacity obscures the underlying mucosa after application, preventing further visualization of the lesion during the procedure. Further studies are required to better define the role of hemostatic powders, establish optimal use settings, and evaluate long-term efficacy and safety in bleeding control.

PuraStat® is a novel gel that provides several advantages over traditional hemostatic powders. Its transparency allows for continuous visualization of the bleeding site, and it can be applied in narrow spaces or in combination with other treatments. The pre-filled syringe design facilitates ease of handling and precise delivery.

To date, most published data on PuraStat® as a haemostatic agent originates from surgical settings. In endoscopy, its primary applications have been in polypectomy-related haemostasis and the promotion of wound healing. Reports indicate a haemostasis success rate of 90.4%, with a recurrence rate of 10.4%. However, data on its efficacy in UGIB lesions remain limited.

This study hypothesizes that PuraStat®, when combined with Adrenaline, represents a feasible and effective first-line treatment for gastrointestinal bleeding, potentially matching or surpassing the current standard of care. A prospective, randomized, parallel-group, open-label clinical trial is proposed. During endoscopy, patients requiring treatment will be randomly assigned to one of two groups: standard care or Adrenaline injection combined with PuraStat®. If haemostasis is not achieved with the initial treatment, the alternative approach will be applied. Patients will be monitored for 30 days to assess bleeding recurrence. The study aims to enroll 126 patients (63 per group).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Undergoing endoscopic therapy for non-variceal gastrointestinal bleeding

Exclusion Criteria:

* Variceal or portal hypertension-related gastrointestinal bleeding
* Lack of signed consent form
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 30 days
  Absence of rebleeding (recurrence of haematemesis, maelena and /or haematochezia, recurrent tachycardia or hypotension after achieving hemodynamic stability, or a reduction in haemoglobin ≥ 2 g/dL after a stable haemoglobin value has been attained) observed within the first 4 weeks following the initial endoscopic treatment.

SECONDARY OUTCOMES:
Technical success | During endoscopy
  Ability to achieve haemostasis and/or complete the endoscopic treatment satisfactorily
Duration of the procedure | During endoscopy
  From the bleeding lesion is detected until the end of the endoscopic treatment.

OTHER OUTCOMES:
Level of difficulty | During endoscopy
  Graded in three categories: Very Easy (no difficulties encountered and no effort needed), Easy (mild difficulties and mild effort needed), Difficult (difficulties encountered and a considerable effort needed or Very Difficult (high difficulties and high effort or skills needed to treat the lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Arnau de Vilanova de Lleida, Lleida, Spain